CLINICAL TRIAL: NCT07169474
Title: Treatment of Peri-trapezial Osteoarthritis With Isolated Trapeziometacarpal Arthroplasty
Brief Title: Treatment of Peritrapezial Osteoarthritis With Isolated Trapeziometacarpal Arthroplasty in 300 Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Benjamin DEGEORGE, Surgeon, Clinique Saint Jean, France
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TM2025
Record Dates: First submitted 2025-08-29; First posted 2025-09-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Trapeziometacarpal Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isolated trapeziometacarpal arthroplasty (Experimental): Isolated TM arthroplasty with double mobility in all cases, using a MAIA (Laboratoire LEPINE) or TOUCH (Laboratoire KERIMEDICAL) prosthesis, depending on the surgeons' habits. Participating surgeons will follow a common operating protocol to ensure consistency of procedures.
  Interventions: Procedure: Isolated trapeziometacarpal arthroplasty with double mobility

INTERVENTIONS:
Procedure: Isolated trapeziometacarpal arthroplasty with double mobility — Isolated trapeziometacarpal arthroplasty with double mobility in all cases, using a MAIA or TOUCH prosthesis depending on the operator's habits.

SUMMARY:
The aim of this clinical trial is to assess the functional outcomes of isolated trapeziometacarpal joint arthroplasty in adult patients requiring surgical management of trapeziometacarpal osteoarthritis, with or without associated symptoms.

The primary endpoint is the evolution of the Quick DASH functional score between inclusion (preoperative) and one year postoperatively.

The study design is a follow-up study of a multicenter cohort.

ELIGIBILITY:
Inclusion Criteria:- Patients over 18 years of age who are members or beneficiaries of french social security

* Patient requiring surgical management
* Clinical and radiographic diagnosis of peri-trapezial osteoarthritis in the 1 or 2 joints:

TM osteoarthritis: glickel sign + grinding test STT osteoarthritis: pain on wrist mobilization in flexion-extension and prono-supination

* TM (Eaton-Littler stages II to III) and STT (Crosby stages II and III) radiographic osteoarthritis
* Persistent pain and functional limitations despite conservative treatment for at least 6 months (combining intermittent immobilization of wrist and thumb + joint infiltration of the 2 joints)
* Ability to understand and sign the informed consent form.

Exclusion Criteria:

* History of surgery on the affected thumb.
* Systemic inflammatory diseases (e.g. rheumatoid arthritis).
* Active infection or history of joint infection of the upper limb.
* Inability to participate in post-operative follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (Quick Dash) functional score | One year
  Change in Quick DASH functional score between inclusion (preoperative) and one year postoperatively, from 0 = no disability to 100 = maximum disability.

SECONDARY OUTCOMES:
Patient satisfaction | 3 months, 6 months and 12 months post-operative
  Likert satisfaction scale at 3 months, 6 months and 12 months post-operative. Chossing between very satisfied , Satisfied , No opinion , Dissatisfied or Very dissatisfied
Complication or surgery | One year
  Need for repeat surgery and any post-operative complication during 12-month follow-up. Need for additional surgery on STT joint (= if pain on palpation and flexion/extension mobilization)
Radiographic evaluation | one year
  Radiographic evaluation: absence of prosthesis complications
Pain in the operated hand | 3 months, 6 months and 12 months postoperatively
  Visual Analogue Scale (VAS) for pain preoperatively at 3 months, 6 months and 12 months postoperatively, from 0 (no pain) to 10 (maximum pain).
Pinch and grip force | 3 months, 6 months and 12 months postoperatively
  Pinch and grip force measured with dynamometer preoperatively, at 3 months, 6 months and 12 months postoperatively.
Range of motion of the thumb | 3 months, 6 months and 12 months postoperatively
  Range of motion of the thumb measured relative to the 2nd metacarpal: antepulsion, retropulsion, abduction and adduction preoperatively, at 3 months, 6 months and 12 months postoperatively
Wrist range of motion | 3 months, 6 months and 12 months postoperatively
  Wrist range of motion: flexion, extension, radial tilt and ulnar tilt preoperatively, at 3 months, 6 months and 12 months postoperatively
Amplitude of possible metacarpophalangeal hyperextension | preoperatively at 3 months, 6 months and 12 months postoperatively
  Amplitude of possible metacarpophalangeal hyperextension preoperatively at 3 months, 6 months and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: benjamin Degeorge, Principal Investigator — Clinique Saint jean sud de france
Locations (1):
- Clinique St jean sud de france, Montpellier, France